CLINICAL TRIAL: NCT00129844
Title: Randomized Phase II Trial of Single Agent Motexafin Gadolinium for Second Line Treatment of Non-Small-Cell Lung Cancer
Brief Title: Study of Motexafin Gadolinium (MGd) for Second Line Treatment of Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0227
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Adenocarcinoma; Non-Small-Cell Lung Carcinoma; Lung Neoplasms
Keywords: Motexafin Gadolinium; non-small cell, lung cancer; Lung cancer; cancer of the lung; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium

SUMMARY:
The purpose of this study is to determine the effect of MGd in non-small-cell lung cancer (NSCLC) when given alone, and to evaluate the difference between two dosing regimens.

DETAILED DESCRIPTION:
Outline:

Two-arm, open-label, randomized, 2-stage Phase II trial. Patients will be randomized on the first stage to 1 of 2 treatment arms:

Arm A - 10 mg/kg MGd once per week

Arm B - 15 mg/kg MGd once every 3 weeks

Patients will be treated on 3 week cycles, up to a maximum of 8 cycles (24 weeks). Patients with either objective response or stable disease after 2 cycles will receive up to 8 cycles of therapy. Patients with progressive disease will be terminated from the study.

At the end of Stage I, both treatment arms will be evaluated, and only the arm(s) that demonstrate at least one response (Complete Response or Partial Response) will proceed to Stage II. If both arms demonstrate a response, then both will proceed to Stage II.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* Histologically or cytologically confirmed diagnosis of NSCLC
* Unresectable locally advanced (Stage IIIB) or metastatic (Stage IV) NSCLC patients who have received one prior platinum-based chemotherapy regimen
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* ECOG performance status score of 0 or 1
* Willing and able to provide written informed consent

Exclusion Criteria:

* Laboratory values of:

  * Absolute neutrophil count < 1500/ul;
  * Platelet count < 75,000/ul;
  * Hemoglobin < 10 gm/dl;
  * AST or ALT > 3 x the upper limit of normal (ULN);
  * Alkaline phosphatase > 5 x ULN;
  * Bilirubin > 2 x ULN;
  * Serum creatinine > 2.0 mg/dL.
* Symptomatic or uncontrolled (untreated or treated and progressing) brain metastasis.
* Evidence of meningeal metastasis.
* Greater than one prior cytotoxic regimen (not counting adjuvant or neoadjuvant cytotoxic chemotherapy if completed > 12 months prior to cytotoxic regimen).
* Chemotherapy, radiation therapy, experimental therapy, immunotherapy or systemic biologic anticancer therapy within 21 days before beginning study treatment.
* Significant weight loss > 10% of body weight in preceding 6 weeks.
* Treatment for another cancer within 3 years of enrollment, unless basal cell carcinoma or cervical cancer in situ.
* Myocardial infarction within 6 months of enrollment or congestive heart failure rated New York Heart Association (NYHA) Class III or IV.
* Uncontrolled hypertension (systolic blood pressure > 160 mm Hg and diastolic blood pressure > 110 mm Hg on maximal medical therapy).
* Known history of porphyria (testing not required at screening visit).
* Known history of glucose-6-phosphate dehydrogenase (G6PD) deficiency (testing not required at screening visit).
* Known history of HIV infection (testing not required at screening visit).
* Female who is pregnant or lactating (serum pregnancy test is required for all female patients of childbearing potential).
* Sexually active male or female of childbearing potential unwilling to use adequate contraceptive protection.
* Physical or mental condition that makes patient unable to complete specified follow-up assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To estimate the response rates of two different MGd dosing regimens for the treatment of NSCLC

SECONDARY OUTCOMES:
To select the most effective regimen based on tumor response
To estimate the time to progression
To estimate survival
To evaluate the safety and tolerability of 2 dosing regimens of MGd in NSCLC patients

CONTACTS AND LOCATIONS:
Overall Officials: Robert Natale, M.D., Study Chair — Aptium Oncology, Inc. Cedars-Sinai Outpatient Cancer Center
Locations (16):
- United States (11):
  - Fountain Valley, California
  - Los Angeles, California
  - Palm Springs, California
  - Columbia, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Rochester, New York
  - Akron, Ohio
  - Knoxville, Tennessee
  - Nashville, Tennessee
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kingston, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec